CLINICAL TRIAL: NCT06254170
Title: Effect of Supplementation With Euterpe Edulis on the Physical and Mental Performance of Healthy Men Subjecting to Physical Exercise
Brief Title: Supplementation Performance And Exercise With Euterpe Edulis for Men's Enhancement
Acronym: SPAEME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Vila Velha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: T015M02-2024MS004; 6.202.888 (Registry Identifier: Plataforma Brasil)
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2023-11

CONDITIONS: Clinical Trial
Keywords: Anti-inflammatory; Antioxidant; Euterpe edulis; Exercise; Juçara
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Euterpe Edulis suplementation (Experimental): Male, aged between 19 and 30 years and practicing physical exercises regularly for at least 3 months will receive the Euterpe Edulis juice for 10 days.
  Interventions: Dietary Supplement: Euterpe Edulis juice; Dietary Supplement: Placebo
- Placebo (Placebo Comparator): Male, aged between 19 and 30 years and practicing physical exercises regularly for at least 3 months will receive the placebo product for 10 days.
  Interventions: Dietary Supplement: Euterpe Edulis juice; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Euterpe Edulis juice — The preparation will be obtained with the same methods already well established in previous studies (SCHULZ et al., 2016.; MENDES et al., 2021). Participants will receive commercial samples of juçara (E.edulis) refrigerated to 4°C to 10°C, per day, for 10 days, and on the 11th will be the exercise and on this day will be administered the juice of the juçara 2 h before on the day of the monitored exercise. The chemical characterization of Euterpe edulis will be with at least 350.0 + or - 17.5 mg of total phenolics (gallic acid equivalent), 186.0 + or - 7.5 mg of total monomeric anthocyanins (cyanidin 3-glycoside), 0.73 + or less 0.01 g of proteins, and 2.75 + or - 0.03 g of lipids (ether extract). During the 10 days of previous treatment, maintain the routine of physical exercises.
  Other Names: Juçara juice
Dietary Supplement: Placebo — Participants will receive 250 ml of water + purple dye + pectin (control) refrigerated to 4°C to 10°C, per day, for 10 days, and on the 11th will be the exercise and on this day will be administered the juice of the juçara 2 h before on the day of the monitored exercise. The chemical characterization of Euterpe edulis will be with at least 350.0 + or - 17.5 mg of total phenolics (gallic acid equivalent), 186.0 + or - 7.5 mg of total monomeric anthocyanins (cyanidin 3-glycoside), 0.73 + or less 0.01 g of proteins, and 2.75 + or - 0.03 g of lipids (ether extract). During the 10 days of previous treatment, maintain the routine of physical exercises.

SUMMARY:
The study aims to evaluate the effect of supplementation with Euterpe edulis on the physical and mental performance, inflammation, muscle recovery, and muscle strength of healthy men submitted to physical exercises. The study will use a double-blind and randomized design, including physical tests, blood sample analysis, and subjective assessments. Participants will receive 250 ml of the juice or a placebo for ten days before the evaluations.

DETAILED DESCRIPTION:
The Euterpe edulis palm, known as juçara, produces spherical and purple fruits, similar to those of the Euterpe oleracea and Euterpe precatoria palms, from where the popular name açaí originates. The juçara fruit has been gaining prominence in the scientific world for its interesting nutritional composition, rich in antioxidants, and for its sustainable production model. Intermittent high-intensity exercise (HIIE) can improve the anti-inflammatory state. Juçara juice (JFJ) has well-established antioxidant and anti-inflammatory properties. Recently, relevant biological activities have been associated with the fruit of the juçara, and its use in food has become an important nutritional, environmental and economic alternative. The objective of this project is to evaluate the antioxidant and anti-inflammatory effects of E. edulis juice after physical exercise in physical activity practitioners. This is a clinical trial, double blind, where high intensity physical exercise will be used and evaluated simple reaction psychomotor test, psychomotor test of choice reaction, collection of blood samples for analysis of interleukins and TNF alpha, strength markers, through the use of dynamometer, jump test, functional tests, muscle endurance test and subjective analysis of fatigue. The selection will be simple random probabilistic according to the inclusion criteria: male gender, aged between 19 and 30 years and practitioners of physical activity for at least 3 months 4 x per week, without comorbidities, non-athlete, non-smokers, and BMI < 30. Participants will receive 250 ml of the juice or placebo during 10 days of previous treatment, maintaining the exercise routine. The aminogram of JFJ (250 ml) will be evaluated to understand the amount of essential amino acids and the possibility of classifying the Juçara fruit as a super fruit. It is expected, after supplementation with the aqueous extract of E. edulis, improvement in the physical and mental capacity of the sample that used the JFJ, in addition to a better response in plasma inflammatory biomarkers and antioxidant capacity, resulting in a positive modulation of the inflammatory profile. In addition, we consider an optimization in muscle recovery capacity and objective and subjective increase in muscle strength as an outcome.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 19 to 30 years, who perform regular physical exercises, in total of 150 min per week, at a minimum of 3 months

Exclusion Criteria:

* Men who use steroids, anabolics, taurine, BCCA, and exogenous supplementation will be excluded.
* People who have motor problems, cardiovascular changes, have type I and II diabetes, smokers, athletes, cognitive deficits, and psychomotor disorders.

Ages: 19 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-19 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Changes in mental capacity - Simple reaction psychomotor test | The test will be applied on day 1 and 11 of the study, after the period of 10 days drinking Juçara juice. The same methodology will be used in the patients who received the placebo product.
  The examined individual should sit in front of the monitor with the index finger of the dominant hand positioned on the sensor (called the ''stand-by key'') located on the control panel. The individual will be instructed to hold their finger on the ''stand-by key'' and move it to the ''reaction key'' as soon as the stimulus (yellow light) appears.
Changes in mental capacity - Psychomotor test of reaction of choice | The test will be applied on day 1 and 11 of the study, after the period of 10 days drinking Juçara juice. The same methodology will be used in the patients who received the placebo product.
  One individual was instructed to respond appropriately and as quickly as possible to stimuli appearing on the screen using the upper and lower limbs.
  Five colored optical stimuli (white, yellow, blue, green, and red) in the form of a circle appeared on the screen, and each circle received its own ''reaction key'' on the control panel that corresponded to the color of the stimulus.
  The examined individual was asked to respond to the stimulus by pressing the corresponding ''reaction key'' with the right or left hand, and the foot was also instructed to press the right or left pedal whenever a white rectangular light appeared on the black background of the screen. Finally, the test included reaction to acoustic stimuli.
Changes in the modulation of the inflammatory profile - Collection of blood samples and analysis of biomarkers | Blood samples will be collected 1 hour before the high-intensity strength exercise and 1 hour after.
  Will be evaluated in the blood samples collected: plasma biomarkers, which include lactate concentration (LA). In plasma, creatine kinase (CK), total antioxidant capacity (TAC) and concentrations of testosterone (T), cortisol © and growth hormone (GH) will be analyzed. In addition to serum concentrations of inflammatory biomarkers such as interleukins (IL-6, IL-8, IL10) and TNF-alpha.
Changes in physical capacity - Dynamometer | The dynamometer will be applied on day 1 and 11 of the study, after the period of 10 days drinking Juçara juice. The same methodology will be used in the patients who received the placebo product.
  The dynamometer is an instrument used to measure muscle strength objectively. In this study will be used the static dynamometer that demonstrated measurement reliability in other clinical trials (HIRANO et al., 2020; MARTINS et al., 2018).
Changes in physical capacity - Jump tests | The jump tests will be applied on day 1 and 11 of the study, after the period of 10 days drinking Juçara juice. The same methodology will be used in the patients who received the placebo product.
  The jump tests are used as a measure of explosive strength and muscle power and this methodology will also be used in this research. The effectiveness of strength assessment in the countermovement jump test has already been validated in other clinical studies (CARBAKAPA et al., 2023).
Changes in physical capacity - Functional tests | The 6-minute step test will be applied on day 1 and 11 of the study, after the period of 10 days drinking Juçara juice. The same methodology will be used in the patients who received the placebo product.
  Functional tests assess strength in more complex movements related to day-to-day activities. In these studies, the 6-minute step test will be applied, as determined its reliability for the evaluation of muscle strength in a previous study (ARCURI et al., 2016).
Changes in physical capacity - Muscular endurance test | The abdominal resistance test will be applied on day 1 and 11 of the study, after the period of 10 days drinking Juçara juice. The same methodology will be used in the patients who received the placebo product.
  Muscle endurance tests assess the ability of muscles to sustain a contraction for a prolonged period. In this study will be used the abdominal resistance test, through the plank test, already reproduced effectively in another study (KOUMANTAKIS et al., 2021).

SECONDARY OUTCOMES:
Subjective change in muscle strength - Subjective analysis of fatigue | The questionnaire will be applied on day 11 of the study, after the period of 10 days drinking Juçara juice and the force tests. The same methodology will be used in the patients who received the placebo product.
  A questionnaire will be developed about the subjective perception of patients about the effects of the treatment employed in the recovery of muscle fatigue. The questions will be based on the Chalder scale and the International Short-Form Physical Activity Questionnaire (IPAQ-SF) (LEE et al., 2011). However, the feeling of improvement or not of physical fatigue after exercise will be the focus of the preparation of a new and unprecedented questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Denise Coutinho Endringer, Study Director — University of Vila Velha

REFERENCES:
- [Background] Arcuri JF, Borghi-Silva A, Labadessa IG, Sentanin AC, Candolo C, Pires Di Lorenzo VA. Validity and Reliability of the 6-Minute Step Test in Healthy Individuals: A Cross-sectional Study. Clin J Sport Med. 2016 Jan;26(1):69-75. doi: 10.1097/JSM.0000000000000190. PMID 25706661
- [Background] Butcher JT, Ali MI, Ma MW, McCarthy CG, Islam BN, Fox LG, Mintz JD, Larion S, Fulton DJ, Stepp DW. Effect of myostatin deletion on cardiac and microvascular function. Physiol Rep. 2017 Dec;5(23):e13525. doi: 10.14814/phy2.13525. PMID 29192067
- [Background] Cabarkapa D, Philipp NM, Cabarkapa DV, Fry AC. Position-specific differences in countermovement vertical jump force-time metrics in professional male basketball players. Front Sports Act Living. 2023 Jul 20;5:1218234. doi: 10.3389/fspor.2023.1218234. eCollection 2023. PMID 37547821
- [Background] Cardoso AL, de Liz S, Rieger DK, Farah ACA, Kunradi Vieira FG, Altenburg de Assis MA, Di Pietro PF. An Update on the Biological Activities of Euterpe edulis (Jucara). Planta Med. 2018 May;84(8):487-499. doi: 10.1055/s-0044-101624. Epub 2018 Feb 21. PMID 29466809
- [Background] Carroll TJ, Taylor JL, Gandevia SC. Recovery of central and peripheral neuromuscular fatigue after exercise. J Appl Physiol (1985). 2017 May 1;122(5):1068-1076. doi: 10.1152/japplphysiol.00775.2016. Epub 2016 Dec 8. PMID 27932676
- [Background] Lee PH, Macfarlane DJ, Lam TH, Stewart SM. Validity of the International Physical Activity Questionnaire Short Form (IPAQ-SF): a systematic review. Int J Behav Nutr Phys Act. 2011 Oct 21;8:115. doi: 10.1186/1479-5868-8-115. PMID 22018588
- [Background] Fang P, She Y, Yu M, Min W, Shang W, Zhang Z. Adipose-Muscle crosstalk in age-related metabolic disorders: The emerging roles of adipo-myokines. Ageing Res Rev. 2023 Feb;84:101829. doi: 10.1016/j.arr.2022.101829. Epub 2022 Dec 20. PMID 36563906
- [Background] Felzenszwalb I, da Costa Marques MR, Mazzei JL, Aiub CA. Toxicological evaluation of Euterpe edulis: a potential superfruit to be considered. Food Chem Toxicol. 2013 Aug;58:536-44. doi: 10.1016/j.fct.2013.05.029. Epub 2013 May 24. PMID 23712094
- [Background] FRANCISCONI, A. F. et al. Genomas completos de cloroplastos e filogenia em três palmeiras Euterpe (E. edulis, E. oleracea e E. precatoria) de diferentes biomas brasileiros. PLoS One, v. 17, n. 7, e0266304, 2022.
- [Background] Hirano M, Katoh M, Gomi M, Arai S. Validity and reliability of isometric knee extension muscle strength measurements using a belt-stabilized hand-held dynamometer: a comparison with the measurement using an isokinetic dynamometer in a sitting posture. J Phys Ther Sci. 2020 Feb;32(2):120-124. doi: 10.1589/jpts.32.120. Epub 2020 Feb 14. PMID 32158074
- [Background] Koumantakis GA, Malkotsis A, Pappas S, Manetta M, Anastopoulos T, Kakouris A, Kiourtsidakis E. Lumbopelvic sagittal standing posture associations with anthropometry, physical activity levels and trunk muscle endurance in healthy adults. Hong Kong Physiother J. 2021 Dec;41(2):127-137. doi: 10.1142/S1013702521500128. Epub 2021 May 4. PMID 34177201
- [Background] Laurindo LF, Barbalho SM, Araujo AC, Guiguer EL, Mondal A, Bachtel G, Bishayee A. Acai (Euterpe oleracea Mart.) in Health and Disease: A Critical Review. Nutrients. 2023 Feb 16;15(4):989. doi: 10.3390/nu15040989. PMID 36839349
- [Background] Martins J, da Silva JR, da Silva MRB, Bevilaqua-Grossi D. Reliability and Validity of the Belt-Stabilized Handheld Dynamometer in Hip- and Knee-Strength Tests. J Athl Train. 2017 Sep;52(9):809-819. doi: 10.4085/1062-6050-52.6.04. Epub 2017 Aug 8. PMID 28787180
- [Background] Martinez Martin A, Perez Herrero M, Sanchez Quiros B, Lopez Herrero R, Ruiz Bueno P, Cocho Crespo S. [Translated article] Benefits of analgesic blocks, PENG block (PEricapsular Nerve Group), in fast recovery after hip surgery. Rev Esp Cir Ortop Traumatol. 2023 Jan-Feb;67(1):T27-T34. doi: 10.1016/j.recot.2022.10.005. Epub 2022 Oct 13. English, Spanish. PMID 36243392
- [Background] Mendes BC, Copetti CLK, Panza VSP, Orssatto LBR, da Rosa JS, Diefenthaeler F, Dalmarco EM, Pietro PFD, Rieger DK. Effects of Euterpe edulis Martius on inflammatory responses to high-intensity intermittent exercise: Crossover randomized trial. Nutrition. 2021 Nov-Dec;91-92:111344. doi: 10.1016/j.nut.2021.111344. Epub 2021 May 28. PMID 34273682
- [Background] de Oliveira AA, Torres AG, Perrone D, Monteiro M. Effect of High Hydrostatic Pressure Processing on the Anthocyanins Content, Antioxidant Activity, Sensorial Acceptance and Stability of Jussara (Euterpe edulis) Juice. Foods. 2021 Sep 22;10(10):2246. doi: 10.3390/foods10102246. PMID 34681295
- [Background] Cunha de Souza Pereira D, Dos Santos Gomes F, Valeriano Tonon R, Beres C, Maria Correa Cabral L. Towards chemical characterization and possible applications of jucara fruit: an approach to remove Euterpe edulis Martius from the extinction list. J Food Sci Technol. 2023 Feb;60(2):429-440. doi: 10.1007/s13197-021-05342-8. Epub 2022 Jan 21. PMID 36712206
- [Background] Petersen AM, Pedersen BK. The anti-inflammatory effect of exercise. J Appl Physiol (1985). 2005 Apr;98(4):1154-62. doi: 10.1152/japplphysiol.00164.2004. PMID 15772055
- [Background] PIETRO, P. F. et al. Efeito do consumo de açaí (Euterpe oleracea Mart.) e de juçara (Euterpe edulis Mart.) sobre biomarcadores metabólicos e de estresse oxidativo em indivíduos saudáveis: um ensaio clínico randomizado cruzado de 4 semanas. Clinical Nutrition, v. 41, n. 1, p. 264-265, 2022.
- [Background] Schulz M, da Silva Campelo Borges G, Gonzaga LV, Oliveira Costa AC, Fett R. Jucara fruit (Euterpe edulis Mart.): Sustainable exploitation of a source of bioactive compounds. Food Res Int. 2016 Nov;89(Pt 1):14-26. doi: 10.1016/j.foodres.2016.07.027. Epub 2016 Aug 3. PMID 28460899
- [Background] Severinsen MCK, Pedersen BK. Muscle-Organ Crosstalk: The Emerging Roles of Myokines. Endocr Rev. 2020 Aug 1;41(4):594-609. doi: 10.1210/endrev/bnaa016. PMID 32393961
- [Background] SHANLEY, P.; MEDINA, G. Frutíferas e plantas úteis na vida amazônica. 1. ed. Belém: Cifor, Imazon, 2005.
- [Background] da Silva W, Machado AS, Souza MA, Mello-Carpes PB, Carpes FP. Effect of green tea extract supplementation on exercise-induced delayed onset muscle soreness and muscular damage. Physiol Behav. 2018 Oct 1;194:77-82. doi: 10.1016/j.physbeh.2018.05.006. Epub 2018 May 7. PMID 29746891
- [Background] Stankiewicz B, Cieslicka M, Mieszkowski J, Kochanowicz A, Niespodzinski B, Szwarc A, Waldzinski T, Reczkowicz J, Piskorska E, Petr M, Skarpanska-Stejnborn A, Antosiewicz J. Effect of Supplementation with Black Chokeberry (Aronia melanocarpa) Extract on Inflammatory Status and Selected Markers of Iron Metabolism in Young Football Players: A Randomized Double-Blind Trial. Nutrients. 2023 Feb 15;15(4):975. doi: 10.3390/nu15040975. PMID 36839333
- [Background] Torre-Villalvazo I, Aleman-Escondrillas G, Valle-Rios R, Noriega LG. Protein intake and amino acid supplementation regulate exercise recovery and performance through the modulation of mTOR, AMPK, FGF21, and immunity. Nutr Res. 2019 Dec;72:1-17. doi: 10.1016/j.nutres.2019.06.006. Epub 2019 Jul 2. PMID 31672317
- [Background] Tutakhail A, Nazari QA, Khabil S, Gardier A, Coudore F. Muscular and mitochondrial effects of long-term fluoxetine treatment in mice, combined with physical endurance exercise on treadmill. Life Sci. 2019 Sep 1;232:116508. doi: 10.1016/j.lfs.2019.05.064. Epub 2019 Jul 3. PMID 31278948
- [Background] Vearrier D, Grundmann O. Clinical Pharmacology, Toxicity, and Abuse Potential of Opioids. J Clin Pharmacol. 2021 Aug;61 Suppl 2:S70-S88. doi: 10.1002/jcph.1923. PMID 34396552
- [Background] Lv Z, Shi W, Zhang Q. Role of Essential Amino Acids in Age-Induced Bone Loss. Int J Mol Sci. 2022 Sep 24;23(19):11281. doi: 10.3390/ijms231911281. PMID 36232583
- See also: IBF - Instituto Brasileiro de florestas. Árvores brasileiras. 2020. Disponível em: https://www.ibflorestas.org.br/lista-de-especies-nativas/palmito-jucara. Acesso em: 5 mai 2023. — https://www.ibflorestas.org.br/lista-de-especies-nativas/palmito-jucara
- See also: IBGE - Instituto Brasileiro de Geografia e Estatística. Censo agropecuário 2017: resultados definitivos. Censo agropecuário. 2017. Disponível em: https://biblioteca.ibge.gov.br/visualizacao/periodicos/3096/agro_2017_resultados_definitivos.pdf. Acesso em: — https://biblioteca.ibge.gov.br/visualizacao/periodicos/3096/agro_2017_resultados_definitivos.pdf

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/70/NCT06254170/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/70/NCT06254170/ICF_001.pdf